CLINICAL TRIAL: NCT05819515
Title: Treatment of Gingival Recession Defects Using Platelet-Rich Fibrin With an Allogenic Dermal Matrix, Compared to the Connective Tissue Graft: A Parallel-arm, Randomized, Controlled, Assessor-blind, Non-inferiority Clinical Trial
Brief Title: Treatment of Gingival Recession Defects Using Platelet-Rich Fibrin With an Allogenic Dermal Matrix
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Hom-Lay Wang, DDS, MSD, Ph D, Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HUM00214311
Record Dates: First submitted 2023-03-21; First posted 2023-04-19 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Connective Tissue Graft (Active Comparator): A connective tissue graft from the patient's palate will be used
  Interventions: Procedure: Tunneled coronally advanced flap
- Allogenic Dermal Matrix with Platelet-Rich Fibrin (Experimental): An allogenic dermal matrix with the patient's platelet-rich fibrin will be used
  Interventions: Procedure: Tunneled coronally advanced flap

INTERVENTIONS:
Procedure: Tunneled coronally advanced flap — Describes the flap design for both treatment arms

SUMMARY:
The study aims to test the non-inferiority of an Allogenic Dermal Matrix with Platelet-Rich Fibrin for treatment of gingival recessions in comparison to the Connective Tissue Graft.

DETAILED DESCRIPTION:
Currently the Connective Tissue Graft (CTG) is referred to as the gold standard in terms of the grafting material for the treatment of gingival recession defects. This study test the non-inferiority of the Allogenic Dermal Matrix (ADM) with Platelet-Rich Fibrin (PRF) to that of the CTG, in terms of the amount of root coverage obtained after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Periodontally and systemically healthy adults
* Full-mouth plaque score and full-mouth bleeding score ≤ 20%
* Presence of at least one 3 mm or deeper gingival recession, with at least 1.5 mm of Keratinized tissue, and 1 mm of gingival thickness) requiring surgical intervention for root coverage
* No interproximal attachment/bone loss
* No prior experience of root coverage procedures within the last 1 year
* The patient must be able to perform good oral hygiene

Exclusion Criteria:

* Contraindications for undergoing periodontal surgery
* Teeth with more than Grade II mobility, or furcation involvement of Class III
* Patients pregnant or attempting to get pregnant (self-reported), or nursing women
* Untreated/active periodontitis, or other untreated acute infections at the surgical site
* Untreated malignancies at the surgical site
* Persistence of uncorrected gingival trauma from traumatic toothbrushing
* Presence of severe tooth malposition, rotation or clinically significant super-eruption
* Self-reported current smoking more than 10 cigarettes/day or pipe or cigar smoking, or active tobacco chewing, or chronic vaping
* Patients with any known history of blood disorders or complications such as abnormal concentration of thrombin and factor XIII in plasma, or hemophilia
* Patients with significant co-morbidities, such as obesity, uncontrolled diabetes, immunosuppression, severe endocrine-induced bone diseases, signs of malnourishment, those receiving immunosuppressive therapy, poor tissue oxygenation or perfusion, and pre- or post-operative radiation
* Patients with known sensitivity to Polysorbate 20, Cefoxitin, Lincomycin, polymyxin B, Vancomycin

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-04-29 (Actual); Primary Completion 2024-03-27 (Actual); Study Completion 2024-03-27 (Actual)

PRIMARY OUTCOMES:
Mean root coverage (mRC) | Assessed at 6 months
  Measured as a percentage of the total baseline recession defect that coverage was obtained at.
Complete root coverage (CRC) | Assessed at 6 months
  Measured as a percentage of total treated sites, that obtained a full coverage of the recession defect
Keratinized tissue (KT) gain | Assessed at 6 months
  Measured in mm
Gingival thickness (GT) gain | Assessed at 6 months
  Measured in mm
Patient-reported outcomes (PROMs) | Measured from the day of the procedure up to a maximum of 1 month
  In terms of pain/discomfort at the palatal donor site or patient's arm. Measured using a scale from 0 (lowest) to 10 (highest).
Duration of surgical procedure | During surgery
  Including the length of surgical procedure, drawing of blood, and preparation of PRF, harvesting of the autogenous CTG. Measured in minutes.

SECONDARY OUTCOMES:
Professionally evaluated esthetic score | Assessed at 6 months
  Assessed using the Root coverage Esthetic Score (RES) system (from 0 lowest, to 10 highest)
Soft tissue volume changes over time | Changes of from baseline (prior to treatment) compared with 3 and 6 months
  Assessed using 3D scanner imaging in the units of mm
Soft tissue volume changes over time | Measured throughout the study to assess changes from immediate post-op (right after the completion of surgical appointment) until the final recall at 6 months
  Assessed using dental ultrasonography in the units of mm
Soft tissue blood flow changes over time | Measured throughout the study to assess changes from immediate post-op (right after the completion of surgical appointment) until the final recall at 6 months
  Assessed and quantified using dental ultrasonography
Patient-reported esthetics | Measured at baseline and at 6 months, and compared between these time points to provide subjective esthetic results
  Based on a visual analogue scale (VAS), measured as numbers from 0 (lowest) to 10 (highest).
Patient-reported satisfaction | Measured at 6 months to provide the satisfaction score in VAS scale
  Based on a visual analogue scale (VAS), measured as numbers from 0 (lowest) to 10 (highest).
Patient-reported post-operative pain as measured with a mobile application | From the day of the procedure until 1 month after the surgical time point
  Measured using a mobile application at the recession grafted site, the donor site on the palate, and the donor site for the venopuncture.

CONTACTS AND LOCATIONS:
Overall Officials: Hom-Lay Wang, DDS MSD PhD, Principal Investigator — University of Michigan; Shayan Barootchi, DMD, MS, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan - Ann Arbor, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Barootchi S, Tavelli L. Tunneled coronally advanced flap for the treatment of isolated gingival recessions with deficient papilla. Int J Esthet Dent. 2022 Feb 17;17(1):14-26. PMID 35175005
- [Background] Barootchi S, Giannobile WV, Tavelli L. PDGF-BB-enriched collagen matrix to treat multiple gingival recessions with the tunneled coronally advanced flap. Clin Adv Periodontics. 2022 Dec;12(4):224-232. doi: 10.1002/cap.10211. Epub 2022 Oct 24. PMID 35665500
- [Background] Tavelli L, Barootchi S. A Minimally Invasive Approach for the Treatment of Multiple Adjacent Gingival Recessions with a Volume-Stable Collagen Matrix: A Case Series. Int J Periodontics Restorative Dent. 2022 Mar-Apr;42(2):155-162. doi: 10.11607/prd.5747. PMID 35353081